CLINICAL TRIAL: NCT01391637
Title: Long-Term Follow-Up Safety and Preliminary Efficacy Study of Human Central Nervous System Stem Cell (HuCNS-SC®) Transplantation in Subjects With Connatal Pelizaeus-Merzbacher Disease (PMD)
Brief Title: Long-Term Follow-Up Study of Human Stem Cells Transplanted in Subjects With Connatal Pelizaeus-Merzbacher Disease (PMD)
Status: Completed | Type: Observational
Sponsor: StemCells, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-N02-PMD
Record Dates: First submitted 2011-07-06; First posted 2011-07-12 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Pelizaeus-Merzbacher Disease; PMD
Keywords: Long term follow-up; HuCNS-SC cells; human central nervous system stem cells
MeSH Terms: conditions — Pelizaeus-Merzbacher Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HuCNS-SC transplanted subjects in the lead-in phase: Subjects who had HuCNS-SC transplant in the lead-in phase study CL-N01-PMD
  Interventions: Biological: HuCNS-SC transplant in the lead-in phase

INTERVENTIONS:
Biological: HuCNS-SC transplant in the lead-in phase — Long-term safety follow-up study

SUMMARY:
The purpose of this study is to determine the long term safety and preliminary effect of HuCNS-SC cells transplanted in subjects with Connatal Pelizaeus-Merzbacher Disease (PMD).

DETAILED DESCRIPTION:
Only subjects who underwent HuCNS-SC transplantation under Protocol CL-N01-PMD will be enrolled in this long term follow-up study.

Subjects will return to the site six months and one year after completion of the Phase I study and then annually for a total study duration of four years. Phone calls will also be made by the Investigator to the subject's parent/legal guardian bi-annually to conduct a phone visit through the four-year duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received HuCNS-SC cells under Protocol CL-N01-PMD

Exclusion Criteria:

* Subjects who received off-protocol immunosuppressive medications.
* Subjects who are concurrently enrolled in another investigational study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PMD Subjects who underwent transplantation of HuCNS-SC cells under CL-N01-PMD study
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse events (SAEs), results of physical and neurological examination, laboratory tests and vital signs. | 4 years

SECONDARY OUTCOMES:
Preliminary efficacy using Bayley-III and Callier-Azusa Scale. | 4 years
  Changes compared to baseline
Changes in brain magnetic resonance imaging (MRI), electroencephalogram (EEG), seizure frequency and somato-sensory evoked potentials (SSEP). | 4 years
  Changes compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Huhn, MD, Study Director — StemCells, Inc.
Locations (1):
- UCSF Medical Center, San Francisco, California, United States